CLINICAL TRIAL: NCT06718751
Title: Tranexamic Acid Therapy For The Treatment of Subdural Hematomas
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Omar Tanweer, Director of Cerebrovascular and Endovascular Neurosurgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-55608
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: tranexamic acid
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PO 650mg TXA tablet (Experimental): 650mg tablets of TXA will be prescribed to be taken orally, once daily for 21 weeks.
  Interventions: Drug: Tranexamic Acid 650 MG
- PO 650mg placebo tablet (Placebo Comparator): 650mg placebo tablet will be prescribed to be taken orally, once daily for 21 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid 650 MG — PO administration of TXA tablet
  Arms: PO 650mg TXA tablet
Drug: Placebo — PO administration of placebo tablet
  Arms: PO 650mg placebo tablet

SUMMARY:
This Phase II randomized, placebo-controlled, double-blinded trial is the first step in our endeavor to improve the clinical outcomes of patients with chronic subdural hematomas (cSDH). Patients who are deemed to not need surgery for their cSDH will be randomly assigned to either the treatment group or the placebo group. Both groups will take a 650mg tablet once daily for 21 weeks and follow the standard of care monitoring for cSDH which is neurological testing and imaging at 6 weeks, 12 weeks, and 21 weeks. With this study, we hope to establish the safety and efficacy of using TXA PO to resolve cSDH without the need for surgical intervention.

DETAILED DESCRIPTION:
Patients must first be evaluated by a neurosurgeon and concluded to be managed conservatively, without a surgical procedure. Then patients may be enrolled into the study if they meet the specific inclusion and exclusion criteria mentioned above.

If the patient signs the informed consent and is enrolled into the study, the treating physician will inform the study team. The patient will be randomized into either treatment or placebo group per the above algorithm. The study will be double-blind, and only the statistician will know the patient groupings.

In the event that unblinding is needed, the statistician will inform the treating physician of the patient's study group.

Tranexamic acid (TXA), the study agent, or matching placebo will be prescribed as a 650mg tablet to be taken once daily for 21 weeks. The drug will be provided as an oral tablet from the pharmacy. The placebo will be a similar tablet. Once prescribed patients will follow the standard of care for conservative management of chronic subdural hematoma.

Baseline evaluation

After obtaining informed consent and prescription of study agent a baseline clinical examination will be done to assess patient's neurological status, including National Institute of Health Stroke Scale (NIHSS), Modified Rankin Score (mRS), and Glasgow Outcome Scale-Extended (GOSE) scales as well as record initial CT scans.

Week 6 follow-up

At the week 6 follow-up, patients will receive a head CT scan to evaluate for changes in hematoma volume and evaluate for coagulopathies. Functional outcomes will also be assessed, including NIHSS, mRS, and GOSE scales.

Week 12 follow-up

At the week 12 follow-up, patients will receive a head CT scan to evaluate for changes in hematoma volume, evaluate for coagulopathies, and hematoma recurrence. Functional outcomes will also be assessed, including NIHSS, mRS, and GOSE scales.

Week 21 follow-up

At the final week 21 follow-up, patients will receive a head CT scan to evaluate for changes in hematoma volume and recurrence. Functional outcomes will also be assessed, including NIHSS, mRS, and GOSE scales.

Standard of care consists of closely monitoring for new neurological symptoms, including altered mental status, focal neurological deficit, headache, or seizures, during hospital admission and during follow-up visits. If new neurological symptoms arise or if existing neurological symptoms do not improve based on progressive or non-resolving hematoma, surgical treatment may be reconsidered. The head CT is part of the standard of care for patients with subdural hematomas. The addition of the study agent, TXA or placebo, is the investigational part of the protocol and not standard of care. Scans will be copied for blinded independent radiologic review, and functional outcomes will be performed by the study physicians.

ELIGIBILITY:
Inclusion Criteria:

* CT scan demonstrating existence of a subdural hematoma, unilateral or bilateral, containing a chronic component
* Neurosurgeon evaluation deemed patient to not need surgery
* Diagnosis within the last 14 days
* Signed informed consent
* Competence to take study medications properly and regularly or access to care giver that is able to comply with accurate study medication administration

Exclusion Criteria:

* Planned surgery, burr-hole craniostomy or mini-craniotomy for their chronic subdural hematoma based on one or more of the following symptoms: medically intractable headache, midline shift >5mm, SDH thickness >10mm, increased ICP, imminent death within 24 hours
* Structural causes for subdural hemorrhage (arachnoid cysts, cortical vascular malformations)
* Recent ischemic stroke
* Other concomitant intracranial pathology (intracranial malignancy)
* Active malignancy
* Need for chronic therapeutic anticoagulation (i.e. atrial fibrillation)
* Acute subdural hematoma with no chronic component
* Active treatment for deep vein thrombosis, pulmonary embolism or cerebral thrombosis (secondary prophylaxis is not considered to be active treatment)
* Known hereditary thrombophilia, including Factor V Leiden, Antithrombin III mutation, Protein C deficiency, Protein S deficiency
* History of thrombosis or thromboembolism, including retinal vein or artery occlusions
* An intrinsic risk of thrombosis or thromboembolism
* Aneurysmal subarachnoid hemorrhage
* Concurrent use of Factor IX complex concentrate or anti-inhibitor coagulant concentrates
* Concurrent use of all-trans retinoic acid
* Active intravascular clotting or disseminated intravascular coagulation
* Need for tissue plasminogen activators
* Known hypersenstivity to TXA or any of the ingredients
* Acute and chronic renal insufficiency indicated by glomerular filtration rate (GFR) < 60 mL/min or creatinine > 2.8 mg/dL
* Hematuria, caused by diseases of renal parenchyma
* Pregnancy or breastfeeding*
* Concomitant hormonal contraception*
* History of convulsions
* History of angioplasty with cardiac stent placement or mechanical heart valve
* Any concern from the attending physician

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Rate of resolution measured as the cSDH volume or diameter | 6 weeks, 12 weeks, 21 weeks

SECONDARY OUTCOMES:
cSDH volume (measured as volume or diameter on follow-up CT scan of the head) | 6 weeks, 12 weeks, 21 weeks
Proportion of patients needing surgery | 12 weeks, 12 weeks, 21 weeks
Hematoma recurrence Hematoma recurrence | 12 weeks, 12 weeks, 21 weeks
Neurological outcome assessed by NIHSS | 6 weeks, 12 weeks, 21 weeks
Functional outcome assessed by mRS | 6 weeks, 12 weeks, 21 weeks
  mRS score is used to assess the degree of disability or dependence in the daily activities of people who have suffered a stroke or other neurological disability
Functional outcome assessed by GOSE | 6 weeks, 12 weeks, 21 weeks
  Glasgow outcome scale extended is a a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery.
Occurrence of adverse events | 6 weeks, 12 weeks, 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omar Tanweer, MD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No